CLINICAL TRIAL: NCT05225493
Title: Supporting Health Care Professionals in Hospital and Primary Care to Promote Adequate HIV Risk and Indicator Condition Driven Testing in Routine Care.
Brief Title: HIV Indicator Diseases in Hospital and Primary Care
Acronym: #AwareHIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Huisartspraktijk Gezondheidscentrum Mathenesserlaan (Unknown); TU Delft department of Artificial Intelligence and MyTomorrows (Unknown); Huisartsen Groep Rotterdam (Unknown); AwareHIV Project Group (Unknown); Huisartspraktijk Handellaan (Unknown); Huisartspraktijk Leerdam (Unknown); Huisartspraktijk Capelle ad IJssel (Unknown); Leiden University Medical Center (Other); Maasstadziekenhuis (Unknown); Rijnstate Hospital (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, Casper Rokx, MD PhD, Erasmus Medical Center
Other Study IDs: MEC-2021-0277
Record Dates: First submitted 2022-01-17; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections; Primary Health Care; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases, Viral; Herpes Zoster; Dermatitis, Seborrheic; Pneumonia; Infectious Mononucleosis; Psoriasis; Candida Infection; Lymphadenopathy; Uterine Cervical Dysplasia; Weight Loss; Diarrhea Chronic; Leukopenia; Thrombocytopenia; AIDS Defining Illness; HIV Indicator Condition
Keywords: General Practitioner, Medical Specialist, HIV indicator condition, HIV risk group, AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases, Viral; Herpes Zoster; Dermatitis, Seborrheic; Pneumonia; Infectious Mononucleosis; Psoriasis; Candidiasis; Lymphadenopathy; Uterine Cervical Dysplasia; Weight Loss; Leukopenia; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital: Medical specialists in hospitals and their patients aged 18 years and older in the participating hospitals who are diagnosed there with an HIV indicator condition.
  Interventions: Behavioral: Peer to peer feedback
- Primary care: General practitioners and their patients aged 18 years and older in the participating general practices who are diagnosed there with an HIV indicator condition.
  Interventions: Behavioral: Peer to peer feedback; Diagnostic Test: HIV rapid test

INTERVENTIONS:
Behavioral: Peer to peer feedback — HIV experts contact non-HIV specialised treating physicians on individual patient care to recommend HIV testing
Diagnostic Test: HIV rapid test — Free HIV rapid tests are provided to non-HIV specialised treating physicians to use in individual patient care in patients at risk of HIV
  Groups: Primary care

SUMMARY:
Patients are frequently evaluated by physicians for medical work-up of HIV indicator conditions in hospital and in primary care at the general practitioner. Testing for HIV is indicated with HIV indicator disorder but often omitted in clinical work-up. Besides the fact that HIV testing is forgotten, there are other reasons such as an underestimation of the risk of HIV in the event of indicator disorders, stigma and difficulties in discussing the test with a patient. Also and more relevant for primary care than for the hospital, practical challenges can exist for a patient to go to a laboratory, or costs are a hurdle.

This project focuses on improving HIV indicator condition driven testing in different settings of the HIV epidemic, initially in the Netherlands as low HIV prevalence setting followed by an assessment of its benefit in different international settings. A specific focus will also be on the Rotterdam area in the Netherlands which has a high prevalence of undiagnosed HIV in the Netherlands. The ultimate aim is to decrease the number of undiagnosed HIV in populations, improve the 90-90-90 HIV cascade of care goals particularly its first pillar, and to help supporting the UNAIDS goal to end HIV/AIDS

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an HIV indicator conditions.

Exclusion Criteria:

* Below 18 years of age
* Recent HIV test (< 12 months, except for mononucleosis-like disease and STDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical specialists, general practitioners and their patients aged 18 years and older in the participating hospitals and primary care who present there with an HIV indicator condition.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The number of adequately performed HIV tests of identified HIV indicator conditions in relation to the total number of identified HIV indicator conditions by physicians in hospital settings during the project. | 3 year
The number of adequately performed HIV tests of identified HIV indicator conditions in relation to the total number of identified HIV indicator conditions by general practitioners in primary care during the project. | 3 year

SECONDARY OUTCOMES:
The number of positive HIV tests in relation to the total number of HIV tests for identified HIV indicator conditions. | 3 year
The percentage of adequately HIV tested patients per HIV indicator condition and per medical specialism. | 31 year
The prevalence of HIV indicator conditions in primary care and hospitals. | 3 year
The incidence of HIV indicator conditions in primary care and hospitals. | 3 year
A sensitive and specific supervised artificial Intelligence tool that recognizes risk factors for HIV and HIV indicator conditions through natural language processing (NLP) and supports the hospital and primary care in proactive HIV testing policies. | 3 year
Acceptance of HIV testing in by patients, medical specialist and in primary care. | 3 year
  Assessed by questionnaire
The costs of pro-active HIV indicator case finding and relation to the savings and QALY's gained | 3 year
  Costs of the program in relation to the savings in costs and QALY's lost as a consequence of earlier HIV diagnosis with subsequent prevented HIV transmission, AIDS comorbidity and hospital admissions.

OTHER OUTCOMES:
The number of HIV tests in relation to the total number of HIV tests done by gender, ethnical background, age, previous HIV test and HIV indicator conditions of the patient, primary care setting and hospital setting. | 3 year
Center for Disease Control and Prevention (CDC) HIV classification of the patients with an HIV positive test. | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Carlijn CCE Jordans, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request

REFERENCES:
- [Derived] Jordans CCE, Niemantsverdriet-Rokx L, Struik JL, van der Waal EC, van der Voorn PVJM, Bakker N, Verbon A, Bindels PJE, Rokx C. Implementing HIV teams to improve HIV indicator condition-guided testing in general practitioner centers in the Netherlands. BMC Prim Care. 2024 Dec 27;25(1):440. doi: 10.1186/s12875-024-02666-0. PMID 39731054